CLINICAL TRIAL: NCT00725296
Title: Remicade Therapy in Psoriatic Arthritis: Investigation of Real Life Regimen in Austria Over 9 Consecutive Infusions
Brief Title: Investigation of 9 Consecutive Infusions of Remicade for Psoriatic Arthritis in Austria (Study P04264)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04264
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remicade (Infliximab): Participants with active and progressive PsA who have responded inadequately to disease-modifying anti-rheumatic drugs will receive induction infusions of Remicade at weeks 0, 2, and 6 given in a dosage due to the decision of the physicians. A maximum of 6 maintenance infusions will be administered with the dosage and interval due to the discretion of the physicians. Whole observation period cannot exceed 102 weeks per participant if the maximal therapy interval of 16 weeks as defined in the Summary of Product Characteristics (SPC) is taken into consideration.
  Interventions: Biological: Remicade (Infliximab)

INTERVENTIONS:
Biological: Remicade (Infliximab) — Induction infusions of Remicade will be administered at weeks 0, 2, and 6 given in a dosage due to the decision of the physicians. A maximum of 6 maintenance infusions will be administered with the dosage and interval due to the discretion of the physicians.
  Other Names: Remicade; SCH 215596

SUMMARY:
This is a prospective, open-label, 1-arm, multicenter observational study to determine the dose and time interval of Remicade (Infliximab) infusions in psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample.

ELIGIBILITY:
Inclusion Criteria:

* Participants with active and progressive psoriatic arthritis who have responded inadequately to disease-modifying anti-rheumatic drugs.

Exclusion Criteria:

* All according to contraindications in the label especially:

  * Participants with tuberculosis or other severe infections such as sepsis, abscesses, and opportunistic infections.
  * Participants with moderate or severe heart failure (NYHA class III/IV).
  * Participants with a history of hypersensitivity to infliximab or to other murine proteins, or to any of the excipients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will receive Remicade induction therapy consisting of 3 infusions in weeks 0, 2, and 6 given in specialized centers. Maintenance therapy will consist of a maximum of 6 infusions given in doses and intervals due to the discretion of physicians.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2004-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 178 participants were enrolled in this study. Of these, 159 participants were Infliximab-naive and 19 participants were already on Remicade (Infliximab). A total of 163 participants received at least one dose: 152 of the 159 naive participants and 11 of the 19 non-naive participants.
Groups:
- Infliximab: Participants with active and progressive psoriatic arthritis (PsA) who have responded inadequately to disease-modifying anti-rheumatic drugs received induction intravenous (IV) infusions of Infliximab at weeks 0, 2, and 6 given in a dosage due to the decision of the physicians and in the usual manner in accordance to the term of the applicable marketing authorization. Then, a maximum of 6 maintenance infusions were administered with the dosage and interval due to the discretion of the physicians. According to the European Summary of Product Characteristics (SPC), Infliximab 5 mg/kg is given as an IV infusion over a 2-hour period followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter.
Period: Overall Study
Arm/Group | Infliximab
Started | 163 (163 of the 178 enrolled participants received at least one dose of Infliximab.)
Completed | 101 (Completed was defined as the number of participants who received 9 consecutive infusions.)
Not Completed | 62
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 3
Not completed — Non-Compliance | 2
Not completed — Lost to Follow-up | 1
Not completed — Other | 38

BASELINE CHARACTERISTICS:
Groups:
- Infliximab: Participants with active and progressive PsA who have responded inadequately to disease-modifying anti-rheumatic drugs received induction intravenous (IV) infusions of Infliximab at weeks 0, 2, and 6 given in a dosage due to the decision of the physicians and in the usual manner in accordance to the term of the applicable marketing authorization. Then, a maximum of 6 maintenance infusions were administered with the dosage and interval due to the discretion of the physicians. According to the European Summary of Product Characteristics (SPC), Infliximab 5 mg/kg is given as an IV infusion over a 2-hour period followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter.
Arm/Group | Infliximab
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of participants was assessed in 163 out of 178 enrolled participants. A total of 163 participants received at least one dose of Infliximab.
  years | 47.96 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Time Interval Between Infusions During Maintenance Therapy
Description: The mean time interval measured in days between Infliximab infusions in participants during the maintenance therapy (between infusion 3/4, 4/5, 5/6, 6/7, 7/8, 8/9) following induction therapy.
Time Frame: Up to 24 months
Population: N= number of Infliximab-naive participants that received induction & maintenance therapy.
  Out of 152 Infliximab-naive participants who were treated, 94 participants received induction therapy (Infliximab at weeks 0, 2, and 6), 83 participants received induction therapy and subsequent maintenance therapy (maximum of 6 maintenance infusions).
Measure: Mean (Standard Deviation); unit: days
Groups:
- Infliximab: Participants with active and progressive psoriatic PsA who have responded inadequately to disease-modifying anti-rheumatic drugs received induction intravenous (IV) infusions of Infliximab at weeks 0, 2, and 6 given in a dosage due to the decision of the physicians and in the usual manner in accordance to the term of the applicable marketing authorization. Then, a maximum of 6 maintenance infusions were administered with the dosage and interval due to the discretion of the physicians. According to the European Summary of Product Characteristics (SPC), Infliximab 5 mg/kg is given as an IV infusion over a 2-hour period followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks thereafter.
Arm/Group | Infliximab
Number analyzed (Participants) | 83
days
  Interval between infusion 3/4 (n= 83) | 57.03 (7.83)
  Interval between infusion 4/5 (n=83) | 57.90 (7.97)
  Interval between infusion 5/6 (n=79) | 58.59 (12.28)
  Interval between infusion 6/7 (n=77) | 56.02 (10.59)
  Interval between infusion 7/8 (n=73) | 56.92 (10.76)
  Interval between infusion 8/9 (n=70) | 59.32 (18.39)

2. Primary Outcome: Median Time Interval Between Infusions During Maintenance Therapy
Description: The median time interval measured in days between Infliximab infusions in participants during the maintenance therapy (between infusion 3/4, 4/5, 5/6, 6/7, 7/8, 8/9) following induction therapy.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Infliximab
Number analyzed (Participants) | 83
days
  Interval between infusion 3/4 (n= 83) | 56 [36 to 84]
  Interval between infusion 4/5 (n=83) | 56 [41 to 84]
  Interval between infusion 5/6 (n=79) | 56 [30 to 114]
  Interval between infusion 6/7 (n=77) | 56 [33 to 115]
  Interval between infusion 7/8 (n=73) | 56 [35 to 119]
  Interval between infusion 8/9 (n=70) | 56 [35 to 159]

3. Primary Outcome: Average Dose During Induction Therapy and Subsequent Maintenance Therapy
Description: The average dose per infusion measured in milligrams/killogram (mg/kg) in participants receiving induction therapy and subsequent maintenance therapy (Infusions 1-3 were induction therapy and infusions 4-9 were maintenance therapy for a total of 9 consecutive infusions).
Time Frame: Up to 24 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Infliximab
Number analyzed (Participants) | 83
mg/kg
  Infusion 1 (n=83) | 3.92 (0.80)
  Infusion 2 (n=83) | 3.92 (0.81)
  Infusion 3 (n=83) | 3.98 (0.86)
  Infusion 4 (n=83) | 3.96 (0.87)
  Infusion 5 (n=83) | 3.94 (0.85)
  Infusion 6 (n=79) | 3.94 (0.85)
  Infusion 7 (n=77) | 3.97 (0.84)
  Infusion 8 (n=73) | 3.97 (0.87)
  Infusion 9 (n=70) | 3.97 (0.89)

4. Primary Outcome: Median Dose During Induction Therapy and Subsequent Maintenance Therapy
Description: The median dose per infusion measured in mg/kg in participants receiving induction therapy and subsequent maintenance therapy (Infusions 1-3 were induction therapy and infusions 4-9 were maintenance therapy for a total of 9 consecutive infusions).
Time Frame: Up to 24 Months
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Infliximab
Number analyzed (Participants) | 83
mg/kg
  Infusion 1 (n=83) | 3.75 [2.70 to 5.71]
  Infusion 2 (n=83) | 3.75 [2.70 to 5.71]
  Infusion 3 (n=83) | 3.75 [2.67 to 5.71]
  Infusion 4 (n=83) | 3.75 [2.67 to 5.71]
  Infusion 5 (n=83) | 3.75 [2.67 to 5.56]
  Infusion 6 (n=79) | 3.75 [2.67 to 5.56]
  Infusion 7 (n=77) | 3.75 [2.67 to 5.56]
  Infusion 8 (n=73) | 3.75 [2.63 to 5.63]
  Infusion 9 (n=70) | 3.75 [2.67 to 5.63]

5. Primary Outcome: Average Overall Dose of All Infusions Per Participant
Description: The average overall dose of all infusions among all Infliximab-naive participants measured in mg/kg.
Time Frame: Up to 24 Months
Population: 152 out of the 159 Infliximab-naive participants were treated in the active phase.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Infliximab
Number analyzed (Participants) | 152
mg/kg | 4.07 (0.84)

6. Primary Outcome: Median Dose of All Infusions Per Participant
Description: The median dose of all infusions among all Infliximab-naive participants measured in mg/kg.
Time Frame: Up to 24 Months
Population: 152 out of the 159 Infliximab-naive participants were treated in the active phase.
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Infliximab
Number analyzed (Participants) | 152
mg/kg | 3.87 [2.53 to 6.41]

ADVERSE EVENTS:
Description: A total of 163 participants out of the 178 enrolled received at least one dose: 152 of the 159 naive participants and 11 of the 19 non-naive participants. Adverse events (AEs) were collected for participants who had received at least one dose of Infliximab.
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 6/163
Other Adverse Events (participants affected / at risk) | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=163)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Demyelinating Polyneuropathy (Nervous system disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No